CLINICAL TRIAL: NCT03252314
Title: Ruptured Aneurysms Treated With Hydrogel Coils
Acronym: RAGE
Status: Active, not recruiting | Type: Observational
Sponsor: Microvention-Terumo, Inc. (Industry)
Collaborators: Semmes-Murphey Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: RAGE
Record Dates: First submitted 2017-08-09; First posted 2017-08-17 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Ruptured Aneurysm
MeSH Terms: conditions — Aneurysm, Ruptured

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Subjects with ruptured aneurysms
  Interventions: Device: Second-generation hydrogel coils

INTERVENTIONS:
Device: Second-generation hydrogel coils — Hydrogel coils 90% by length
  Other Names: HydroFrame; HydroFill; HydroSoft; HydroSoft 3D

SUMMARY:
To determine safety and occlusion rates when second-generation hydrogel coils are used in the treatment of ruptured intracranial aneurysms.

DETAILED DESCRIPTION:
RAGE is a prospective, non-randomized, multicenter, post-market study. The RAGE study is designed to determine the safety and occlusion rates of hydrogel coils in the ruptured aneurysm study population. Secondary objectives include determining clinical outcomes, packing density, occlusion stability, rates of recurrence, rebleed, retreatment, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 18 and ≤ 80 years of age.
2. Patient has a previously untreated, ruptured saccular intracranial aneurysm 2 - 15 mm in diameter for which the clinical decision to treat with hydrogel coil embolization has been made independent of the decision to participate in the study described in this protocol.
3. Patient has a baseline Hunt and Hess Score of I, II, or III.
4. Patient or patient's legally authorized representative has provided written informed consent.
5. Patient must be considered by the treating physician to be available for and able to complete all followup visits.
6. Patient has not been previously entered into this study.

Exclusion Criteria:

1. Inability to obtain written informed consent.
2. Patient is < 18 or > 80 years of age.
3. Patient has a baseline Hunt and Hess score of IV or V.
4. Target aneurysm is dissecting, fusiform, mycotic, blister-like, tumoral, or AVM-related.
5. Target aneurysm maximum diameter is > 15 mm or < 2 mm.
6. Target aneurysm was previously treated via clipping or coiling.
7. Target aneurysm is deemed by the treating physician to be unsuitable for coiling or unlikely to be successfully treated by endovascular techniques.
8. Target aneurysm has not been confidently determined by the treating physician to be the source of SAH.
9. Planned use of a flow diverter or intrasaccular device as a component of the target aneurysm treatment plan.
10. Intended use of a coil-assist stent as a component of the target aneurysm treatment plan, unless use of a stent is 1) planned as a subsequent stage of a staged coiling procedure or 2) used for bailout purposes.
11. Patient has a known, untreatable hypersensitivity to contrast dye, iodine, hydrogel, or any other component of the treatment device.
12. Patient has a contraindication to heparin or aspirin.
13. Patient has vascular anatomy/tortuosity preventing access to the target aneurysm.
14. Patient is unable to undergo DSA or DSA is determined unsuitable or outside standard of care by the treating physician.
15. Patient has a serious or life-threatening comorbidity that could confound study results.
16. Patient is at high risk of noncompliance due to a history of substance abuse, psychosocial issues, etc.
17. Patient is unable to complete scheduled followup assessments due to comorbidities, geographical limitations, or a life expectancy of less than 18 months.
18. Patient is pregnant, breastfeeding, or plans to become pregnant prior to completion of followup.
19. Patient is enrolled in another device or drug study in which participation could confound study results.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 - 80 years with a ruptured saccular intracranial aneurysm in whom coil embolization is determined to be the appropriate treatment strategy.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-11-27 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Death or major stroke | 30 days
Major ipsilateral stroke, neurological death, or rebleeding from the target aneurysm | 18 months
Adequate angiographic occlusion (as defined by the Raymond Roy Occlusion Classification) without interim retreatment secondary to aneurysm recurrence or rebleed of the target aneurysm | 18 months

SECONDARY OUTCOMES:
Rebleed rate of the target aneurysm | 30 days
Rebleed rate of the target aneurysm | 18 months
Modified Rankin Score (mRS) | 18 months
Modified Rankin Score (mRS) | 30 days
Packing density measured by volumetric filling of the aneurysm | Immediately following procedure
Retreatment rate | 18 months
Retreatment rate due to recurrence | 18 months
Adequate angiographic occlusion (as defined by the Raymond Roy Occlusion Classification) without rebleed of the target aneurysm | 18 months
Adequate angiographic occlusion (as defined by the Raymond Roy Occlusion Classification) without rebleed of the target aneurysm or retreatment for residual aneurysm | 18 months
Occlusion Stability (as defined by the Raymond Roy Occlusion Classification) | 18 months
Adverse events related to the device and/or the procedure | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Adam S Arthur, MD, MPH, FACS, Principal Investigator — Semmes-Murphey Clinic; David Fiorella, MD, PhD, Principal Investigator — Stony Brook Medical Center
Locations (1):
- Methodist University Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided